CLINICAL TRIAL: NCT00075400
Title: A Phase II Evaluation of Gleevec(TM) (NCI-Supplied Agent: STI571 [Imatinib Mesylate], NSC# 716051) in the Treatment of Recurrent or Persistent Carcinosarcoma of the Uterus
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent or Persistent Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00653; NCI-2014-00653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000346361; GOG-0230C (Other: Gynecologic Oncology Group); GOG-0230C (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive imatinib mesylate PO QD or BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II clinical trial studies the side effects and how well imatinib mesylate works in treating patients with uterine cancer that has failed to respond to initial chemotherapy or has re-grown after therapy. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the activity of Gleevec^trademark (TM) (imatinib mesylate) as measured by progression-free survival at six months.

II. To determine the frequency and severity of adverse effects of Gleevec^TM in this cohort of patients as assessed by the Common Terminology Criteria of Adverse Events version 3.0 (CTCAE v3.0).

SECONDARY OBJECTIVES:

I. To determine the distribution of progression-free survival and overall survival.

II. To estimate the objective response rate (partial and complete response as defined under the Response Evaluation Criteria In Solid Tumors [RECIST] criteria).

III. To determine the effects of prognostic factors such as initial performance status and histological grade.

TERTIARY OBJECTIVES:

I. To determine the levels of expression of v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (c-KIT), platelet-derived growth factor receptor (PDGFR), v-akt murine thymoma viral oncogene homolog 2 (AKT2), and phosphorylated (p)-AKT2 in archived, formalin-fixed, paraffin-embedded primary tumors collected prior to the initiation of first-line chemotherapy

OUTLINE:

Patients receive imatinib mesylate orally (PO) once daily (QD) or twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed uterine carcinosarcoma that is persistent or recurrent with documented disease progression after appropriate local therapy; acceptable histologic type is defined as carcinosarcoma (malignant mixed Mullerian tumor), homologous or heterologous type
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST; tumors within a previously irradiated field will be designated as "non-target" lesions
* Patients must not be eligible for a higher priority Gynecological Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of carcinosarcoma; initial treatment may include high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
  * Note: Patients on this non-cytotoxic study are allowed to receive one additional cytotoxic chemotherapy regimen for management of recurrent or persistent disease, as defined above; however, due to the novel nature of biologic compounds, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
* Patients must have NOT received any non-cytotoxic chemotherapy for management of recurrent or persistent disease
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to CTCAE v3.0 grade 1
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v3.0 grade 1
* Bilirubin less than or equal to 1.5 x ULN (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE v3.0 grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients who have met the pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception, and cannot be lactating; since interactions with the metabolism of oral contraceptives cannot be excluded, a barrier method of contraception must be used
* Patients must have tissue blocks from initial diagnosis available for submission to the GOG Tissue Bank

Exclusion Criteria:

* Patients who had previous treatment with Gleevec^TM
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Patients with signs or symptoms of bowel dysfunction or obstruction
* Patients receiving therapeutic anticoagulation with warfarin
* Patients with deep venous or arterial thrombosis (including pulmonary embolism) within six weeks of study entry
* Patients receiving therapeutic corticosteroids
* Patients with active or uncontrolled infection
* History of seizures or those patients receiving phenytoin, phenobarbital, or carbamazepine
* Patients with other severe concurrent disease, which the investigator feels may make the patients inappropriate for study entry
* Presence of clinically apparent central nervous system metastases, or other carcinomatous meningitis
* History of myocardial infarction within previous six months or congestive heart failure requiring therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warner Huh, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 1/5/2004 and closed to accrual on 8/1/2005.
Groups:
- Gleevec: Gleevec™ 600 mg QD po continuously (a cycle will be defined as 28 days). If first cycle of Gleevec™ at 600 mg QD is tolerated without any significant toxicity, the dose can be escalated to 400 mg BID po Q 12 hours until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Gleevec
Started | 26
Completed | 23 (Eligible and treated patients.)
Not Completed | 3
Not completed — Ineligible: wrong primary | 1
Not completed — Never treated | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | Gleevec
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.2)
Age, Customized [Number; unit: participants]
  40-49 years | 3
  50-59 years | 3
  60-69 years | 11
  70-79 years | 4
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
FIGO (International Federation of Gynecology and Obstetrics) Stage Recurrent/Persistent [Number; unit: participants] | 23
Histologic Type [Number; unit: participants]
  Carcinosarcoma-homologous | 3
  Carcinosarcoma-heterologous | 8
  Carcinosarcoma, Malignant Mixed Mullerian Tumor | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) > 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: For those patients whose disease can be evaluated by physical examination, progression was assessed prior to each 28-day cycle. CT scan or MRI if used to follow measurable disease every other cycle for the first 6 months.
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Gleevec
Number analyzed (Participants) | 23
percentage of participants | 4.3 [0.2 to 19.0]

2. Primary Outcome: Incidence of Adverse Effects as Assessed by CTCAE v 3.0
Description: The frequency and severity of all toxicities are tabulated from submitted case report forms and summarized for review.
Time Frame: Each cycle during treatment and 30 days after treatment ends.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23
Participants
  Leukopenia | 21 | 2 | 0 | 0 | 0
  Neutropenia | 21 | 1 | 1 | 0 | 0
  Anemia | 7 | 7 | 9 | 0 | 0
  Allergy | 22 | 0 | 1 | 0 | 0
  Hearing | 22 | 0 | 1 | 0 | 0
  Cardiovascular | 22 | 1 | 0 | 0 | 0
  Constitutional | 7 | 9 | 6 | 1 | 0
  Dermatologic | 19 | 3 | 1 | 0 | 0
  Endocrine | 21 | 1 | 1 | 0 | 0
  Gastrointestinal | 5 | 5 | 12 | 1 | 0
  Genitourinary | 22 | 0 | 0 | 1 | 0
  Hemorrhage | 22 | 0 | 1 | 0 | 0
  Lymphatics | 17 | 3 | 2 | 1 | 0
  Metabolic | 18 | 2 | 1 | 1 | 1
  Neuropathy | 21 | 2 | 0 | 0 | 0
  Other neurologic | 21 | 0 | 2 | 0 | 0
  Ocular | 21 | 1 | 0 | 1 | 0
  Pain | 19 | 2 | 2 | 0 | 0
  Pulmonary | 22 | 1 | 0 | 0 | 0
  Sexual | 22 | 1 | 0 | 0 | 0

3. Secondary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; up to 5 years
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Gleevec
Number analyzed (Participants) | 23
percentage of participants | 0 [0.0 to 9.5]

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gleevec
Number analyzed (Participants) | 23
months | 4.1 [3.3 to 8.6]

5. Secondary Outcome: Duration of Progression Free Survival
Description: as for outcome 1
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; up to 5 years
Population: Eligible and treated patients.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Gleevec
Number analyzed (Participants) | 23
months | 1.6099 [0.9199 to 2.1027]

6. Secondary Outcome: Initial Performance Status
Description: Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance Status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work Performance Status 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Gleevec
Number analyzed (Participants) | 23
Participants
  Performance status 0 | 12
  Performance status 1 | 10
  Performance status 2 | 1

7. Secondary Outcome: Initial Histologic Grade
Description: G1 - Highly differentiated adenomatous carcinoma. G2 - Differentiated adenomatous carcinoma with partly solid areas. G3 - Predominantly solid or entirely undifferentiated carcinoma. Not graded - tumor grade not reported.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Gleevec
Number analyzed (Participants) | 23
Participants
  Grade 1 | 0
  Grade 2 | 4
  Grade 3 | 18
  Not graded | 1

8. Other Pre Specified Outcome: PDGFR Expression Levels in Archived, Formalin-fixed, Paraffin-embedded Primary Tumor Tissue by IHC
Description: Potential associations with clinical or PFS response will be assessed.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: AKT2 Expression Levels in Archived, Formalin-fixed, Paraffin-embedded Primary Tumor Tissue by IHC
Description: Potential associations with clinical or PFS response will be assessed.
Time Frame: Baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: p-AKT2 Expression Levels in Archived, Formalin-fixed, Paraffin-embedded Primary Tumor Tissue
Description: Potential associations with clinical or PFS response will be assessed.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: c-KIT Expression Levels in Archived, Formalin-fixed, Paraffin-embedded Primary Tumor Tissue by Immunohistochemistry (IHC)
Description: Potential associations with clinical or PFS response will be assessed.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment
Arm/Group | Gleevec
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gleevec (N=23)
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Death No Ctcae Term - Death Nos (General disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gleevec (N=23)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Rhinitis (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Neutrophils (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 19
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 1
Weight Gain (General disorders) | 1
Fever (General disorders) | 1
Weight Loss (General disorders) | 1
Fatigue (General disorders) | 17
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Flushing (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 4
Distention (Gastrointestinal disorders) | 2
Taste Alteration (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Anorexia (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 8
Hemorrhage, Gu - Vagina (Vascular disorders) | 4
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 1
Liver Dysfunction (Hepatobiliary disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 6
Edema: Head And Neck (Blood and lymphatic system disorders) | 5
Ast (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Neuropathy-Sensory (Nervous system disorders) | 4
Neuropathy-Motor (Nervous system disorders) | 1
Watery Eye (Eye disorders) | 1
Blurred Vision (Eye disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Head/Headache (General disorders) | 4
Pain: Extremity-Limb (General disorders) | 2
Pain: Back (General disorders) | 2
Pain: Abdominal Pain Nos (General disorders) | 3
Pain: Tumor (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Urinary Retention (Renal and urinary disorders) | 2
Incontinence, Urinary (Renal and urinary disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less